CLINICAL TRIAL: NCT03619096
Title: Clinical Comparison Between Two Surgical Techniques for the Treatment of Multiple Gingival Recessions With Porcine Collagen Matrix
Brief Title: Two Different Surgical Techniques for the Treatment of Multiple Gingival Recessions With Porcine Collagen Matrix
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Arthur Belem Novaes Jr, Teacher of Periodontia- Department of Buco Maxillofacial Surgery and Traumatology and Periodontics, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE:65396417000005419
Record Dates: First submitted 2018-01-17; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Gingival Recession; Xenograft Model; Gingival Recession, Generalized
Keywords: Gingival recession; porcine collagen matrix; multiple gingival recessions; tunnel technique
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Split Mouth clinical trial, comparing two different techniques. One side, the tunnel technique will be performed and on the other side, extended flap will be performed. Both surgical techniques will use Porcine Collagen Matrix.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants and the outcomes Assessor are masked about the surgical technique that was performed. The surgical technique ir randomized in accordance with the arch side of each patient, so the investigator will open a envelope just before starting the incisions to know which technique will be performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (tunnel technique) (Active Comparator): It Will be performed root coverage of multiple recessions using porcine collagen matrix with a tunnel Technique
  Interventions: Procedure: tunnel technique for Root coverage with Porcine collagen Matrix
- Control Group (extended flap technique) (Placebo Comparator): It Will be performed root coverage of multiple recessions using porcine collagen matrix with a extended flap technique
  Interventions: Procedure: extended fla technique for Root coverage with Porcine collagen Matrix

INTERVENTIONS:
Procedure: tunnel technique for Root coverage with Porcine collagen Matrix — Tunnel technique for root coverage for multiple gingival recessions, using porcine collagen matrix
  Other Names: mucograft matrix
  Arms: Test Group (tunnel technique)
Procedure: extended fla technique for Root coverage with Porcine collagen Matrix — Extended flap technique for root coverage for multiple gingival recessions, using porcine collagen matrix
  Other Names: mucograft matrix
  Arms: Control Group (extended flap technique)

SUMMARY:
The gold standard for gingival recession treatment is the coronal repositioning of the flap associated with the subepithelial connective tissue graft. The porcine collagen matrix (PCR) has been used as a substitute for subepithelial connective tissue graft in periodontal plastic surgery and has achieved similar results. The PCR use has the advantage of avoiding possible pre and postoperative complications , as well as overcome the limitations presented by autograft . The different surgical techniques used for root coverage seek predictability and success . For this, besides the type of incision placements flap and graft are the most important because the healing benefits and outcome .

The aim of this study is to compare two surgical techniques for root coverage and evaluate which one provides better clinical outcomes and less morbidity . 20 adults , nonsmoking patients , showing multiple bilateral gingival recessions , class I or II Miller located in canine, first and second premolars are selected. Both techniques use the PCR as a graft . However, in one Quadrant partial flap will be held together with relaxing incisions through an intrasulcular incision, PCR will be positioned 1 mm apical to the cementoenamel junction (CEJ) and the flap will be positioned 1 mm coronal CEJ. In the opposite quadrant periosteal envelope that does not use relaxing incisions, avoiding any scars, will be performed with the PCR. The clinical parameters (gingival recession height and width, keratinized tissue thickness and width) will be evaluated 2 weeks after basic periodontal therapy and after 6 and 12 months to surgical procedures..

ELIGIBILITY:
Inclusion Criteria:

-bilateral multiple gingival recession type Miller class I or II with at least one tooth with 3 mm of gingival recession height

Exclusion Criteria:

* diabetics
* pregnant women
* chronic use of medication
* periodontitis
* smokers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2019-07-06 (Estimated)

PRIMARY OUTCOMES:
Root coverage (milimeters) | baseline, 6 and 12 motnhs
  Root Coverage is measured by the difference between Gingival Recession Hight at baseline and 12 months

SECONDARY OUTCOMES:
Keratinized tissue (milimeters) | baseline, 6 and 12 months
  Keratinized tissue is measured by its width and thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Belem Novaes JR, Principal Investigator — University of Sao Paulo
Locations (1):
- Marilia Bianchini Lemos Reis, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided